CLINICAL TRIAL: NCT01076595
Title: Prospective Multicenter, Non Interventional Study to Evaluate the Patient's Characteristics Associated With Adherence to Treatment Regimen by Betaferon in the BetaPlus Program
Brief Title: Prospective, Multicenter Non Interventional Study to Evaluate Adherence to Betaferon Over a 2 Years Period
Acronym: SEPLUS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15098; BF0910FR (Other: company internal)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; BetaPlus program; Recurrent/remittent multiple sclerosis patients; Adherence to treatment regimen
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Betaferon 250 microgram

SUMMARY:
The aim of the SEPLUS study is to evaluate the patients characteristics associated with adherence to Betaferon over a 24-month follow up period after the initiation of Betaferon in the BetaPlus program

ELIGIBILITY:
Inclusion Criteria:

* Male or female >/= 18 years old
* Outpatient with a confirmed diagnosis of Recurrent-Remittent multiple sclerosis or patients at high risk of developing multiple sclerosis after a first demyelinating clinical event
* Patient who initiated Betaferon as described by SmPC less than 2 months ago. The decision of physician is clearly separated from the decision to include the patient in the study
* Treatment naïve patients before the initiation of Betaferon
* OR Patients having interrupted Betaferon for more than 6 months before to start again
* OR Patients receiving a disease modifying drug (DMD) other than Betaferon
* Patient with EDSS score < 4
* Patients approved and signed an inform consent and approved the collect of their data

Exclusion Criteria:

* Contraindications and warning of the respective Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2010-05; Primary Completion 2013-11 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The adherence to treatment (rate of patients continuing with Betaferon® regimen after 24 months) | 24 months

SECONDARY OUTCOMES:
Compliance to Betaferon according physician (rate of patients with compliance rater > 94,5%) | 6 months, 12 months, 24 months
Adherence to treatment (rate of patients continuing with the Betaferon® regimen at 6 and 12 months) | 6 months, 12 months
Rate of patients with prematurely study discontinuation | 0-6 months, 6-12 months, 12-18 months, 18-24 months
Patient's autonomy with regard to the Betaferon® injections (Number of injections realized by the patient alone/total number of injections) | 24 months
Tolerability of Betaferon injections (rate and number of injections) | 24 months
Patient's Quality of Life (Mean total score of FAMS [Functional Assessment of Multiple Sclerosis]) | 24 months
Fatigue (mean total score of FSS [Fatigue Severity scale]) | 24 months
Progression of clinical Condition( annual rate of Relapses) | 24 months
Percentage of patients with change of in EDSS (Expanded Disability Status Scale) < 1 between M0 and end of the study | 24 months
Percentage of patients with change in EDSS< 1 and no relapse between M0 and M24 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, France